CLINICAL TRIAL: NCT06286501
Title: Identification of Adolescent Patients at Risk of Oral Diseases and Targeting of Preventive Treatment, and the Use of Antibacterial Photodynamic Therapy as an Adjunctive Treatment Method
Brief Title: Targeting of Preventive Treatment for Adolescents at Risk of Oral Diseases
Acronym: LumoPrevent
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wellbeing Services County of Pirkanmaa (Other)
Collaborators: Tampere University (Other); University of Helsinki (Other); Metropolia University of Applied Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R23060L
Record Dates: First submitted 2024-02-22; First posted 2024-02-29 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Dental Caries in Children; Dental Plaque; Tooth Decay; Periodontitis
Keywords: Antibacterial; Preventive oral care; Lumoral
MeSH Terms: conditions — Dental Plaque; Dental Caries; Periodontitis

STUDY DESIGN:
Intervention Model Description: Randomized clinical study on a CE-approved medical device
Who Masked: Outcomes Assessor
Masking Description: Data will be collected using individual study codes for participants. Study codes do not reveal which group the participant has belonged to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): Standard, personalized oral hygiene and Lumoral Treatment home-use
  Interventions: Device: Lumoral Treatment; Other: Standard, personalized oral health care
- Control group (Active Comparator): Standard, personalized oral hygiene
  Interventions: Other: Standard, personalized oral health care

INTERVENTIONS:
Device: Lumoral Treatment — Home-use photodynamic antibacterial dual-light oral health care device with a marker substance
  Arms: Study group
Other: Standard, personalized oral health care — Home-based oral health care instructed by a professional, with emphasis on personal needs according to oral condition and previous oral health care habits.

SUMMARY:
The aim of the study is to identify adolescent patients that are at risk of developing oral diseases, and to assess if targeted preventive oral treatment with antibacterial dual-light therapy as an adjunctive treatment method can have a positive impact in preventing oral diseases from emerging.

DETAILED DESCRIPTION:
Good oral health is an essential factor in people's general and psychosocial well-being. According to the Global Burden of Disease 2020, untreated dental caries (tooth decay) in permanent teeth is the most common health condition. Modern dietary habits in developed countries, with increased consumption of sugar and other products that are known to have a negative impact on oral health need to be looked at both at regional and global levels. Educational programs that promote oral health awareness and emphasize the importance of good oral hygiene may be effective in encouraging adolescents to adopt healthy habits.

Globally, tooth decay is very common among children (WHO 2022), and in Finland, the oral health of children and adolescents has deteriorated in recent years. However, the risk of a young person's tooth decay can be reduced by promoting good oral hygiene by implementing less destructive dietary habits and enhanced oral health habits.

Poor dental plaque control causes increased oral bacterial burden, which is known to be associated with inflammatory oral diseases, such as periodontitis. Periodontitis is very common in Finland, for example, according to a national Health 2000 survey, the prevalence was 64 % in the adult population, and 10-15 % in adolescents. Periodontitis can lead to tooth loss, and there is a link between periodontitis and many systemic diseases as untreated periodontitis may maintain low-grade inflammation in the body.

Recent studies have identified effective methods, such as the aMMP-8 point-of-care test, for identifying oral inflammatory burden, also on adolescents. New tools in fighting a global battle against bacteria-caused tooth decay are welcome. Antibacterial photodynamic therapy (aPDT) and antibacterial blue light (aBL) have emerged as solutions for attacking dental biofilm. Until recently, these treatment methods have only been available in an office setting. A group of Finnish scientists has developed a new and unique home-use aPDT and aBL method, which has proven to have a very strong emphasis on eliminating harmful oral bacteria. The method is used along with the best-so-far home-based dental care, brushing, and flossing.

ELIGIBILITY:
Inclusion Criteria:

* 14-16 years old, and a junior high school 8th-grade pupil from the area of the Wellbeing Services of County Pirkanmaa
* Agreement to participate in the study and to sign a written consent form, including either consent from caregiver(s) with pupils under 14 years, or information to caregiver(s) with pupils from 15 to 16 years old
* Able to cooperate with the treatment

Exclusion Criteria:

* Presence of any physical limitation or restriction that might restrict Lumoral use
* Unwilling to participate in the study
* Periodontal treatment within 3 months prior to study

Ages: 14 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2024-04-18 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Bleeding on probing (BOP) | 12 months
  Change in bleeding on probing (BOP)
  A full-mouth assessment at six sites per tooth (mesiobuccal, buccal, distobuccal, mesiolingual, lingual, distolingual) Gingival bleeding is considered as positive if bleeding occurs within 15 seconds after gentle probing with a probe at the sulcus Dichotomous scoring to each site of the tooth as bleeding "1 present" and "0 absent" BOP is reported as the percentage (%) of sites with positive findings Calculation formula: number of bleeding sites/ 6 times number of teeth.
Bleeding on probing (BOP) | 6 months
  Change in bleeding on probing (BOP)
  A full-mouth assessment at six sites per tooth (mesiobuccal, buccal, distobuccal, mesiolingual, lingual, distolingual) Gingival bleeding is considered as positive if bleeding occurs within 15 seconds after gentle probing with a probe at the sulcus Dichotomous scoring to each site of the tooth as bleeding "1 present" and "0 absent" BOP is reported as the percentage (%) of sites with positive findings Calculation formula: number of bleeding sites/ 6 times number of teeth.

SECONDARY OUTCOMES:
Active matrix metalloproteinase 8 (aMMP-8) | 12 months
  Change in the accurate periodontal inflammation marker aMMP-8 level at 12 months compared to baseline.
  The aMMP-8 marker analysis will be performed using Periosafe chairside test (Dentognostics GmbH) according to the manufacturer's instructions.
Probing Pocket Depth (PPD) | 6 months
  Change in the Probing Pocket Depth (PPD)
  A full-mouth assessment, measured at 4 sites per tooth Assessed from the base of the pocket to the gingival margin (mm)
Probing Pocket Depth (PPD) | 12 months
  Change in the Probing Pocket Depth (PPD)
  A full-mouth assessment, measured at 4 sites per tooth Assessed from the base of the pocket to the gingival margin (mm)
Visible plaque index (VPI) | 6 months
  Change in VPI
  * Assessment of six index teeth, measured at four sites per tooth
  * Dichotomous scoring to each site of the tooth as plaque "1 present" and "0 absent"
  * VPI reported as the percentage (%) of sites with plaque
  * Calculation formula: number of sites with plaque/ 4 times number of teeth.
Visible plaque index (VPI) | 12 months
  Change in VPI
  * Assessment of six index teeth, measured at four sites per tooth
  * Dichotomous scoring to each site of the tooth as plaque "1 present" and "0 absent"
  * VPI reported as the percentage (%) of sites with plaque
  * Calculation formula: number of sites with plaque/ 4 times number of teeth.
Decayed tooth assessment (DT) | 12 months
  Change in the number of decayed teeth.
  A full-mouth examination, the number of untreated decayed permanent teeth will be calculated.
Clinical attachment level (CAL) | 6 months
  Change in CAL.
  A full mouth assessment. CAL is a combination of two measurements: 1) at least 2 mm distance from the gingival margin to the cementoenamel junction (CEJ ), and 2) probing depth. The calculation (x + x) forms the CAL value.
Clinical attachment level (CAL) | 12 months
  Change in CAL.
  A full mouth assessment. CAL is a combination of two measurements: 1) at least 2 mm distance from the gingival margin to the cementoenamel junction (CEJ ), and 2) probing depth. The calculation (x + x) forms the CAL value.
Microbiological evaluation/16S rRNA analysis | 6 months
  Change in composition of bacterial flora at 12 months compared to the baseline.
  A microbial sample shall be obtained from a periodontal pocket, or from the Cementoenamel junction using a paper point. Quantification of periodontopathic bacteria by 16S rRNA sequencing analysis.
  - Microbiological samples can be collected using Iso Taper Paper Points, size-20 (VDW GmbH) from selected gingival/periodontal pockets with maximum initial probing depth. The paper points can be placed into sterile, small-aliquot containers, and immediately stored at -20°C until analysis
Microbiological evaluation/16S rRNA analysis | 12 months
  Change in composition of bacterial flora at 12 months compared to the baseline.
  A microbial sample shall be obtained from a periodontal pocket, or from the Cementoenamel junction using a paper point. Quantification of periodontopathic bacteria by 16S rRNA sequencing analysis.
  - Microbiological samples can be collected using Iso Taper Paper Points, size-20 (VDW GmbH) from selected gingival/periodontal pockets with maximum initial probing depth. The paper points can be placed into sterile, small-aliquot containers, and immediately stored at -20°C until analysis
Oral-related quality of life measurement (OHIP-14) | 12 months
  OHIP-14 is a standardized questionnaire for oral-related symptoms. It measures people's perception of the social impact of oral disorders on their well-being.
  Fourteen items of OHIP are divided into seven dimensions: functional limitation, physical discomfort, psychological discomfort, physical disability, psychological disability, social disability, and handicaps. (Slade GD 1997). Responses are made on a 5-point scale (from 0 = never, to 4 = very often).
Absence of adverse effects | 12 months
  The presence of device-related serious adverse events (SAE) or any patterns of device-related adverse events (AE) will be monitored and the number of incidents will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Maria Heikkinen, Professor, Principal Investigator — Wellbeing Services of County Pirkanmaa
Locations (1):
- Wellbeing Services of County Pirkanmaa, Tampere, Pirkanmaa, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] GBD 2017 Oral Disorders Collaborators; Bernabe E, Marcenes W, Hernandez CR, Bailey J, Abreu LG, Alipour V, Amini S, Arabloo J, Arefi Z, Arora A, Ayanore MA, Barnighausen TW, Bijani A, Cho DY, Chu DT, Crowe CS, Demoz GT, Demsie DG, Dibaji Forooshani ZS, Du M, El Tantawi M, Fischer F, Folayan MO, Futran ND, Geramo YCD, Haj-Mirzaian A, Hariyani N, Hasanzadeh A, Hassanipour S, Hay SI, Hole MK, Hostiuc S, Ilic MD, James SL, Kalhor R, Kemmer L, Keramati M, Khader YS, Kisa S, Kisa A, Koyanagi A, Lalloo R, Le Nguyen Q, London SD, Manohar ND, Massenburg BB, Mathur MR, Meles HG, Mestrovic T, Mohammadian-Hafshejani A, Mohammadpourhodki R, Mokdad AH, Morrison SD, Nazari J, Nguyen TH, Nguyen CT, Nixon MR, Olagunju TO, Pakshir K, Pathak M, Rabiee N, Rafiei A, Ramezanzadeh K, Rios-Blancas MJ, Roro EM, Sabour S, Samy AM, Sawhney M, Schwendicke F, Shaahmadi F, Shaikh MA, Stein C, Tovani-Palone MR, Tran BX, Unnikrishnan B, Vu GT, Vukovic A, Warouw TSS, Zaidi Z, Zhang ZJ, Kassebaum NJ. Global, Regional, and National Levels and Trends in Burden of Oral Conditions from 1990 to 2017: A Systematic Analysis for the Global Burden of Disease 2017 Study. J Dent Res. 2020 Apr;99(4):362-373. doi: 10.1177/0022034520908533. Epub 2020 Mar 2. PMID 32122215
- [Background] Aytac Bal F, Ozkocak I, Cadirci BH, Sirin Karaarslan E, Cakdinleyen M, Agaccioglu M. Effects of photodynamic therapy with indocyanine green on Streptococcus mutans biofilm. Photodiagnosis Photodyn Ther. 2019 Jun;26:229-234. doi: 10.1016/j.pdpdt.2019.04.005. Epub 2019 Apr 6. PMID 30965147
- [Background] Chapple IL, Bouchard P, Cagetti MG, Campus G, Carra MC, Cocco F, Nibali L, Hujoel P, Laine ML, Lingstrom P, Manton DJ, Montero E, Pitts N, Range H, Schlueter N, Teughels W, Twetman S, Van Loveren C, Van der Weijden F, Vieira AR, Schulte AG. Interaction of lifestyle, behaviour or systemic diseases with dental caries and periodontal diseases: consensus report of group 2 of the joint EFP/ORCA workshop on the boundaries between caries and periodontal diseases. J Clin Periodontol. 2017 Mar;44 Suppl 18:S39-S51. doi: 10.1111/jcpe.12685. PMID 28266114
- [Background] Costa SA, Nascimento GG, Colins PMG, Alves CMC, Thomaz EBAF, Carvalho Souza SF, da Silva AAM, Ribeiro CCC. Investigating oral and systemic pathways between unhealthy and healthy dietary patterns to periodontitis in adolescents: A population-based study. J Clin Periodontol. 2022 Jun;49(6):580-590. doi: 10.1111/jcpe.13625. Epub 2022 Apr 19. PMID 35415936
- [Background] Dimenas SL, Jonsson B, Andersson JS, Lundgren J, Petzold M, Abrahamsson I, Abrahamsson KH. A person-centred, theory-based, behavioural intervention programme for improved oral hygiene in adolescents: A randomized clinical field study. J Clin Periodontol. 2022 Apr;49(4):378-387. doi: 10.1111/jcpe.13601. Epub 2022 Feb 23. PMID 35132653
- [Background] Heikkinen AM, Raivisto T, Raisanen I, Tervahartiala T, Bostanci N, Sorsa T. Implementing of aMMP-8 point-of-care test with a modified new disease classification in Finnish adolescent cohorts. Clin Exp Dent Res. 2022 Oct;8(5):1142-1148. doi: 10.1002/cre2.603. Epub 2022 Jun 8. PMID 35676762
- [Background] Hentila J, Laakamaa N, Sorsa T, Meurman J, Valimaa H, Nikinmaa S, Kankuri E, Tauriainen T, Patila T. Dual-Light Photodynamic Therapy Effectively Eliminates Streptococcus Oralis Biofilms. J Pharm Pharm Sci. 2021;24:484-487. doi: 10.18433/jpps32084. PMID 34559627
- [Background] Nikinmaa S, Moilanen N, Sorsa T, Rantala J, Alapulli H, Kotiranta A, Auvinen P, Kankuri E, Meurman JH, Patila T. Indocyanine Green-Assisted and LED-Light-Activated Antibacterial Photodynamic Therapy Reduces Dental Plaque. Dent J (Basel). 2021 May 3;9(5):52. doi: 10.3390/dj9050052. PMID 34063662
- [Background] Pussinen PJ, Paju S, Viikari J, Salminen A, Taittonen L, Laitinen T, Burgner D, Kahonen M, Lehtimaki T, Hutri-Kahonen N, Raitakari O, Juonala M. Childhood Oral Infections Associate with Adulthood Metabolic Syndrome: A Longitudinal Cohort Study. J Dent Res. 2020 Sep;99(10):1165-1173. doi: 10.1177/0022034520929271. Epub 2020 Jun 1. PMID 32479136
- [Background] Pakarinen S, Saarela RKT, Valimaa H, Heikkinen AM, Kankuri E, Noponen M, Alapulli H, Tervahartiala T, Raisanen IT, Sorsa T, Patila T. Home-Applied Dual-Light Photodynamic Therapy in the Treatment of Stable Chronic Periodontitis (HOPE-CP)-Three-Month Interim Results. Dent J (Basel). 2022 Nov 2;10(11):206. doi: 10.3390/dj10110206. PMID 36354651
- [Background] Raisanen IT, Sorsa T, Tervahartiala T, Raivisto T, Heikkinen AM. Low association between bleeding on probing propensity and the salivary aMMP-8 levels in adolescents with gingivitis and stage I periodontitis. J Periodontal Res. 2021 Apr;56(2):289-297. doi: 10.1111/jre.12817. Epub 2020 Dec 11. PMID 33305834
- See also: Heikkinen, AM. Oral health, smoking and adolescence. Doctoral dissertation. University of Helsinki, Faculty of Medicine. Nov 2011. — http://urn.fi/URN:ISBN:978-952-10-7250-5
- See also: Aromaa, A, Koskinen S. Health and functional capacity in Finland : Baseline results of the Health 2000 health examination survey. National Public Health Institute. 2004. — https://urn.fi/URN:NBN:fi-fe201204193452
- See also: Honkala S, (ed.), Heikka H, (ed.), Heikkinen M, (ed.), Helenius-Hietala J, (ed.), Sirviö K, (ed.). Terve suu. Helsinki: Kustannusosakeyhtiö Duodecim, 2020. 464 p. — https://researchportal.helsinki.fi/en/publications/terve-suu
- See also: Periodontitis ("Gum disease"). Duodecim current care guidelines. May 2018. — https://www.kaypahoito.fi/xmedia/hoi/khp00096_engl.pdf
- See also: Raivisto T, Sorsa T, Räisänen IT, Kauppila T, Ruokonen H, Tervahartiala T, Haukka J, Heikkinen AM.Active Matrix Metalloproteinase-8 Chair Side Mouth Rinse Test, Health Behaviour and Oral Health in Finnish Adolescent Cohort.J Clin of Diagn Res.2020. — http://dx.doi.org/10.7860/JCDR/2020/43031.13467
- See also: WHO - Oral Health. World Health Organization Newsroom, March 2023. — https://www.who.int/news-room/fact-sheets/detail/oral-health